CLINICAL TRIAL: NCT01727453
Title: Randomized Controlled Trial to Compare Treatment With Oral Anticoagulation With Antagonists of vitaminK vs Low Molecular Weight Heparin(Bemiparin) in Patients With Anticoagulation Criteria and an Episode of Gastrointestinal Bleeding.
Brief Title: Compare VKA vs LMWH in Patients With Anticoagulation Criteria and Episode of Gastrointestinal Bleeding.
Acronym: HEPACO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPACO
Record Dates: First submitted 2012-10-31; First posted 2012-11-16 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Acute Gastrointestinal Bleeding
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bemiparin (Active Comparator): Group 1 (low molecular weight heparin: bemiparin), which is the study group: after passing the bleeding episode, will receive low molecular weight heparin (bemiparin) in anticoagulant dose. Check should be made by measurement of anti-factor Xa.
  Interventions: Drug: Bemiparina
- Warfarin (Active Comparator): which is the control group will receive VKA anticoagulation as before they had the bleeding episode, with regular monitoring by measurement of prothrombin time (INR). Patients taking acenocoumarol before bleeding episode will be treated with warfarin and the once who were receiving warfarin will continue with the same treatment. Treatment control is performed by measuring the INR periodically.
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: warfarin — Warfarin in anticoagulant dose
  Other Names: VKA oral anticoagulationin
  Arms: Warfarin
Drug: Bemiparina — Group 2 (VKA oral anticoagulation: warfarin), which is the control group will receive VKA anticoagulation as before they had the bleeding episode, with regular monitoring by measurement of prothrombin time (INR). Patients taking acenocoumarol before bleeding episode will be treated with warfarin and the once who were receiving warfarin will continue with the same treatment. Treatment control is performed by measuring the INR periodically.
  Randomization will be performed using sealed opaque envelopes that contain the treatment option that will be obtained through a list of random numbers generated by computer.
  Arms: Bemiparin

SUMMARY:
SUMMARY

1.0. Type of Application: Clinical trial comparing two treatments in terms of authorized use.

1.1. Promoter: Institute of Research, Hospital de la Santa Creu i Sant Pau. Avgda. Sant Antoni M.Claret, 167. 08025 Barcelona. Tel: (34) 93 291 9140/93 291 21 73.

1.2. Title: Randomized controlled trial to compare treatment with oral anticoagulation with antagonists of vitamin K versus low molecular weight heparin (Bemiparin) in patients with anticoagulation criteria and who have had an episode of gastrointestinal bleeding.

1.3. Protocol code: HEPACO 1.4. Principal Investigators: Dr. Candid Villanueva Sanchez. Dr. Jose Mateo Arranz. Contributors: Dr. Alicia Brotons (Service of Digestive Pathology), Dr. Angela Puente (service of Digestive Pathology), Dr. Isabel Graupera (Service of Digestive Pathology) and Dr. Marina Carrasco (Hematology Service). Hospital de la Santa Creu i Sant Pau. Avgda. Sant Antoni Maria Claret, 167. 08025 Barcelona. Tel: (34) 93 291 91 39. Fax: (34) 93 291 92 78.

E-mail: cvillanueva@santpau.es. 1.5. Centers that are planned for the trial: Service Gastroenterology and Hematology Service of the Sant Creu i Sant Pau, Barcelona.

1.6. Clinical Research Ethics Committee: Hospital de la Santa Creu i Sant Pau. 1.7. Monitor: Institute for Research (CAIBER) of the Hospital de Sant Pau. Avgda. Sant Antoni M.Claret, 167. 08025 Barcelona. Tel: (34) 93 291 9140.

1.8. Drugs: warfarin, bemiparin. 1.9. Development stage: Clinical Trial phase IV 1.10. Main objective: To compare the incidence of gastrointestinal rebleeding and safety of oral anticoagulation versus low molecular weight heparin in patients who have had an acute gastrointestinal bleeding and have indication for anticoagulation.

1.11. Design: prospective open clinical trial, randomized and controlled. 1.12. Study disease: acute gastrointestinal bleeding. 1.13. Primary endpoint of the valoration: Incidence of gastrointestinal bleeding.

1.14. Study population and total number of patients: 20 patients were required in each group (40 total) to objectify a decrease of rebleeding rate of 45% with an alpha error of 5% and 10% beta.

1.15. Treatment duration: 2 years. 1.16. Calendar and expected completion date: July 2011 - July 2013

DETAILED DESCRIPTION:
4.c. OBJECTIVES: The main objective of this prospective, randomized study is to evaluate whether the substitution of VKA therapy for low molecular weight heparin (bemiparin) in patients who have had an episode of gastrointestinal bleeding and have the indication for anticoagulant therapy, is associated with a decreased incidence of recurrent gastrointestinal bleeding.

Secondary objectives consist of all of the following:

* Incidence of thromboembolic events
* Bleeding from other locations
* Severity of recurrent episodes of haemorrhagea
* Transfusion requirements
* Identification of risk factors associated
* Mortality

  5. TYPE OF TRIAL AND DESING.

This is a prospective, randomized, controlled trial, in which patients with gastrointestinal bleeding and indication for anticoagulation will be randomized into two treatment groups:

Group 1 (low molecular weight heparin: bemiparin), which is the study group: after passing the bleeding episode, will receive low molecular weight heparin (bemiparin) in anticoagulant dose. Check should be made by measurement of anti-factor Xa.

Group 2 (VKA oral anticoagulation: warfarin), which is the control group will receive VKA anticoagulation as before they had the bleeding episode, with regular monitoring by measurement of prothrombin time (INR). Patients taking acenocoumarol before bleeding episode will be treated with warfarin and the once who were receiving warfarin will continue with the same treatment. Treatment control is performed by measuring the INR periodically.

Randomization will be performed using sealed opaque envelopes that contain the treatment option that will be obtained through a list of random numbers generated by computer.

6. SELECTION OF SUBJECTS 6.1 CRITERIA FOR INCLUSION AND EXCLUSION:

6.1.1. Inclusion criteria: patients with anticoagulant treatment criteria (treated with acenocoumarol or warfarin) and high or very high risk of embolism, who have an acute gastrointestinal bleeding (high or low) endoscopically untreatable, secondary to multiple vascular lesions, diverticular origin or unclarified origin (after VGC and DC) who have no exclusion criteria.

6.1.2. Exclusion criteria. Not be included patients with one or more of the following criteria: A) less than 18 years old. B) pregnancy. C) patient refusal to participate in the study. D) patients in whom the decision has been taken not to provide active treatment for the existence of any clinical situation considered terminal (severe associated diseases evolved).

E) Contraindication LMWH (allergy, heparin induced thrombocytopenia). F) bleeding secondary to esophageal varices and / or gastric. G) associated bleeding peptic injury. H) bleeding secondary to tumors or polyps. i) Presence of portal hypertension with or without cirrhosis. J) bleeding due to Mallory-Weiss syndrome. K) anticoagulation for low risk embolic lesions.

6.2 DIAGNOSTIC CRITERIA AND DEFINITIONS:

* Acute upper gastrointestinal bleeding: presence of hematemesis and / or melena noted by the medical staff. Any acute gastrointestinal bleeding episode is defined as the presence of macroscopic signs of bleeding (hematemesis, rectal bleeding, hematochezia and / or melena) noted by the medical staff. Severe gastrointestinal bleeding is defined as one that also present hemodynamic repercusion (systolic blood pressure <100 mm Hg and heart rate> 100 bpm) or hemoglobin (Hb) <80 g / l decrease in Hb> 20 g / l in 24 hours.
* Upper GI bleeding caused by peptic ulcer, in which cases urgent endoscopy identify an ulcer with one of the following stigmata of recent haemorrhage: 1) active arterial bleeding jet or oozing hemorrhage2) non-bleeding visible vessel, 3) clot attached, 4) indirect signs of bleeding (spots deep ulcer), and 5) ulcer without signs and evidence of blood remains in the gastric lumen without other potentially bleeding lesions.
* Variceal hemorrhage, those cases where urgent endoscopy identify varices with one of the following signs of bleeding: 1) active bleeding or oozing /spurting, 2) adherent clot on varices or platelet clot, with recent blood remnants in esophagogastric light, or 3) varices with red blood in esophagogastric light in the absence of other injuries in complete endoscopic examination.
* Upper GI bleeding non-variceal neither ulceral origin, those cases where urgent endoscopy identifies a lesion (Mallory-Weiss, Dieulafoy lesion, angiodysplasia or other), with active bleeding, non-bleeding visible vessel, or adherent clot.
* Lower gastrointestinal bleeding, those cases with evidence of bleeding (melena or hematochezia), in which urgent endoscopy is normal and has no history of hematemesis or coffee ground vomiting.
* Rebleeding hemorrhage cases that present 1) new hematemesis or recurrence/ persistence of fresh melena, associate with 2) a decrease in hemoglobin greater than 20 g / l in a period of less than 24 hours, or hemodynamic (TAS <100 mmHg and / or heart rate> 100 ppm). All cases will be assessed through a new emergency endoscopy to confirm it is a recurrence and proceed to a second endoscopic treatment if it's necessary.
* Very high thromboembolic risk:

  1. Patients in the first month after they have had an episode of venous thromboembolism.
  2. Presence of mitral or tricuspid mechanical valve.
  3. Multiple mechanical prostheses.
* High risk of thromboembolism, any mechanical prosthesis (except mitral or tricuspid that they are very high risk), atrial fibrillation embolism, valvular atrial fibrillation, venous thromboembolism in the first three months or thrombophilia, atrial fibrillation at high risk (index CHA2DS2- VASC ≥ 4, see table in appendix).
* Low thromboembolic risk: atrial fibrillation (CHA2DS2-VASC index <4), venous thromboembolism more than 6 months.
* Mortality: Any death that occurs during the course of the study. We considered attributable to bleeding all deaths within 30 days after clinical onset of bleeding, whatever the immediate cause of death.

  7. DESCRIPTION OF TREATMENT. Initially, hemodynamic stabilization shall be of all patients according to clinical practice.

During the bleeding episode prophylactic dose heparin will be administered by continuous infusion (120 mg / d 1-2mg/kg/d), starting at 6 hours after the administration of vitamin K. After 48 hours without clinical signs of hemorrhagic activity (with no macroscopic blood remnants) will start the treatment of choice (at thehospital). Patients randomized to VKA receive will warfarin. Patients receiving acenocoumarol will take warfarin. Patients randomized to receive LMWH will receive bemiparina (Hibor) to maintain an a-Xa levels between 0.4-1.0 U / ml.

8. ASSAY DEVELOPMENT AND EVALUATION OF RESPONSE. 8.A. Parameters to evaluate: The following primary and secondary parameters were evaluated:

1. Primary variables: incidence of upper or lower gastrointestinal bleeding in the follow-up period in both groups. Acute gastrointestinal bleeding it will be recorded, when they occur, at any time during the monitoring period. Is defined as any acute gastrointestinal bleeding episode in which medical care personnel finds the presence of macroscopic signs of bleeding (hematemesis, rectal bleeding, hematochezia and / or melena). Serious Gastrointestinal bleeding is defined as one that also present hemodynamic repercussion (systolic blood pressure <100 mm Hg and heart rate> 100 bpm) or hemoglobin (Hb) <80 g / l decrease in Hb> 20 g / l in 24 hours.
2. Secondary variables:

2.1-Mortality: We included all deaths in this period whatever the reason immediately. Shall specify the date of death to calculate the actuarial probability curves. This will be considered as time 0, the entry in the first hospital where the patient go, or the first bleeding sign if the patient were hospitalized.

where and when they were admitted first symptom of bleeding. 2.2-Severity of rebleeding (TA, FC, low Hb, transfusion requirements). 2.3- Association with NSAIDs, aspirin or other antiplatelet agents. 2.5 -treatment complications. It will collect any adverse events observed during follow-up, either initially or not attributable to treatment. Notification of serious adverse events and unexpected will be modeled and general instructions contained in Royal Decree 223/2004 of 6 February laying down the requirements for conducting clinical drug trials 2.6-Time of hospitalization during follow-up. 2.7-Number of hospitalizations during follow-up. 2.8-In case of rebleeding, is reported: initial anticoagulation level, endoscopic findings, endoscopic treatment, etc.

8.B.Study development:

* Initially there will be an evaluation of all patients with anticoagulation criteria (treated with acenocoumarol or warfarin) that present and upper or lower gastrointestinal bleeding. All patients were submit to an initial clinical evaluation including history and physical examination and request a blood test (with blood count, biochemistry and coagulation), ECG, chest radiography and abdominal ultrasonography. Anticoagulation be corrected by the administration of vitamin K (10 mg) and analytical control are performed at 6 hours to check the reversal of the anticoagulation.
* Then it will be a diagnosis or therapeutic endoscopy as early as possible (at least partial correction of anticoagulation, INR <1.6). All patients will be practised VGC (also in patients with suspected lower gastrointestinal bleeding, to rule out completely high origin). In patients with lower gastrointestinal bleeding (normal VGC), after conducting VGC will be VCC. In cases where the source of bleeding is not clarified with gastroscopy and colonoscopy, capsule endoscopy was carried out, and according to its results shall be practised an enteroscopy (forward/backward or both). Furthermore it will practised an endoscopy, only if the clinical situation of each case requires. In both groups, all suspected rebleeding be evaluated by endoscopy.
* As mentioned in point 7, during the bleeding episode will be administered to all patients prophylactic dose heparin and after 48 hours without clinical signs of hemorrhagic activity it will be divided the participation in the study and proceed to randomization for treatment LMWH vs. warfarin.
* Once the acute episode is resolved, outpatient will be visited at 30th day and then every 3 months (complete blood counts).
* Controls of anticoagulant therapy using anti-Xa or INR it will be held every four weeks, except in the cases that need to change the dose, in which cases the controls will be more frequent.

ELIGIBILITY:
Inclusion Criteria:patients with anticoagulant treatment criteria (treated with acenocoumarol or warfarin) and high or very high risk of embolism, who have an acute gastrointestinal bleeding (high or low) endoscopically untreatable, secondary to multiple vascular lesions, diverticular origin or unclarified origin (after VGC and DC) who have no exclusion criteria.

-

Exclusion Criteria:Not be included patients with one or more of the following criteria:

A) less than 18 years old. B) pregnancy. C) patient refusal to participate in the study. D) patients in whom the decision has been taken not to provide active treatment for the existence of any clinical situation considered terminal (severe associated diseases evolved).

E) Contraindication LMWH (allergy, heparin induced thrombocytopenia). F) bleeding secondary to esophageal varices and / or gastric. G) associated bleeding peptic injury. H) bleeding secondary to tumors or polyps. i) Presence of portal hypertension with or without cirrhosis. J) bleeding due to Mallory-Weiss syndrome. K) anticoagulation for low risk embolic lesions

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Rebleeding | 1 year
  upper or lower gastrointestinal bleeding in the follow-up period in both groups.

SECONDARY OUTCOMES:
thromboembolic events | 1 year
Mortality: | 1 year
  We included all deaths in this period whatever the reason immediately. Shall specify the date of death to calculate the actuarial probability curves. This will be considered as time 0, the entry in the first hospital where the patient go, or the first bleeding sign if the patient were hospitalized.
  where and when they were admitted first symptom of bleeding.
Severity of rebleeding | 1 year
  TA, FC, low Hb, transfusion requirements).
Association with NSAIDs, aspirin or other antiplatelet agents. | 1 year
treatment complications. | 1 year
  It will collect any adverse events observed during follow-up, either initially or not attributable to treatment. Notification of serious adverse events and unexpected will be modeled and general instructions contained in Royal Decree 223/2004 of 6 February laying down the requirements for conducting clinical drug trials
Time of hospitalization | 1 year
  Time of hospitalization during follow-up.
Number of hospitalizations during follow-up. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Candido Villanueva, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain